CLINICAL TRIAL: NCT04085471
Title: CTHRC1 Apromising Biomarker in Rheumatoid Arthritis Diagnosis
Brief Title: CTHRC1 Abiomarker in Rheumatoid Arthritis Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lobna Amer Araby Ahmed, Principal investigator, Assiut University
Other Study IDs: rheumatoid arthritis
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CTHRC1 biomarker level in rheumatoid arthritis — measurment of levels of CTHRC1 in patients diagnosed as RA

SUMMARY:
The purpose of the study is to determine whether plasma levels of the collagen triple helix repeat containing (CTHRC1) protein can serve as a blood-based biomarker for diagnosis of rheumatoid arthritis (RA) ,and furthermore its correlation with disease activity.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, progressive, autoimmune disease of synovial joints. Characterized by periods of flares with high disease activity involving both a systemic immune response and tissue-specific inflammatory events that can lead to erosive joint and bone destruction and subsequent disability . Currently, diagnosis of RA is based mainly on the extent of tenderness and swelling of the joints , levels of acute-phase reactants such as C-reactive protein (CRP) ,erythrocyte sedimentation rate(ESR) , high titers of rheumatoid factor (RF) and high titers of antibodies against cyclic citrullinated peptide (anti-CCP) in the plasma .Of interest, CTHRC1 is a secreted modulator of Wnt signaling, which is a key regulator of joint remodeling, and promotes cell proliferation and migration. Therefore, CTHRC1 may contribute to multiple aspects of the pathogenic FLS behavior in RA and modulate processes that promote synovial hyperplasia and invasion.The expression pattern of CTHRC1 in pannus, its role in the function of FLS relevant to cartilage damage in RA, and CTHRC1's association with disease severity in murine arthritis raised the question of whether CTHRC1 could be used as a marker for RA diagnosis and monitoring of disease activity in patients

ELIGIBILITY:
Inclusion Criteria:

* -Patients diagnosed as RA.
* Patients ( >18)who are age and sex matched with the controls

Exclusion Criteria:

. Other Rheumatologic diseases. .Patients with malignancy . .Patients with hepatic disease .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: measurement of CTHRC1in RA patints
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
CTHRC1 Apromising biomarker in rheumatoid arthritis diagnosis | one year
  measurement of levels of CTHRC1 in rheumatoid arthritis patients

REFERENCES:
- [Background] Myatt GL, Ecobichon DJ, Greenhalgh R. Fenitrooxon and S-methyl fenitrothion: acute toxicity and hydrolysis in mammals. Environ Res. 1975 Dec;10(3):407-14. doi: 10.1016/0013-9351(75)90036-5. No abstract available. PMID 2462